CLINICAL TRIAL: NCT01452516
Title: A Prospective, Multi-Center, Nonrandomized Study to Assess Lumbar Fusion Using Interbody Cages With Autograft in Conjunction With Instrumented Posterolateral Gutter Fusions Using NanOss Bioactive
Brief Title: Effectiveness of Lumbar Fusion When NanOss Bioactive Is Used With Posterolateral Gutter Fusions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated due to slow accrual rate.
Sponsor: Pioneer Surgical Technology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B01-2010
Record Dates: First submitted 2011-09-02; First posted 2011-10-17 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-11

CONDITIONS: Degenerative Disc Disease; Spinal Stenosis; Spondylolisthesis
Keywords: PLF; lumbar fusion; bone graft; biologics
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nanOss Bioactive Bone void filler (Other): Lumbar fusion using interbody cages with autograft in conjunction with instrumented posterolateral gutter fusions using nanOss Bioactive bone void filler
  Interventions: Device: nanOss Bioactive Bone void filler; Device: Interbody FCage

INTERVENTIONS:
Device: nanOss Bioactive Bone void filler — Instrumented posterolateral gutter fusions using nanOss Bioactive bone void filler
Device: Interbody FCage — Lumbar fusion using interbody cages with autograft. This will be done in conjunction with the posterolatreal gutter fusion

SUMMARY:
Spine fusion is one of the most common procedures performed in spinal surgery. Several surgical techniques can achieve a solid union, but the intertransverse posterolateral fusion (PLF) is the most widely used. However, complications can develop when the bone graft material used is insufficient to achieve the desired fusion. With its unique properties, nanOss Bioactive can be mixed with bone marrow aspirate (BMA) and other graft materials to obtain new bone growth during the healing process.

It is hypothesized that the use of nanOss Bioactive will result in fusion at 12 months, with CT evidence of bridging trabecular bone, less than 3mm of translational motion, and less than 5 degrees of angular motion. In addition, patients are expected to see an improvement in Oswestry Disability Index scores, VAS pain scores, and SF36 scores, while decreasing the use of pain medication, returning to work, and finding satisfaction in the results of their surgery.

DETAILED DESCRIPTION:
The post marketing clinical trial is designed to assess lumbar fusion using interbody cages with autograft in conjunction with instrumented posterolateral gutter fusions using nanOss Bioactive bone void filler in patients with degenerative disc disease (DDD) characterized by the inclusion and exclusion criteria listed below.

Patients for this study will be recruited from up to 10 clinical sites. It is estimated that 100 patients will be enrolled in the study. At least 10 investigators will participate in the study. Patients who meet the inclusion and exclusion criteria will be asked to sign the informed consent. Preoperatively, the patient will provide his /her medical history and complete self assessment forms. The investigator will perform a clinical evaluation.

Patients who meet the criteria for entrance into the study will undergo lumbar fusion using interbody cages with autograft in conjunction with instrumented posterolateral gutter fusions using nanOss Bioactive in combination with local autograft and bone marrow aspirate (BMA). Anterior lumbar interbody fusion procedures are not allowed.

Following surgery, operative and discharge information will be collected. The patients will be evaluated at 6 weeks, 6 months and 12 months postoperatively. At each postoperative visit, the investigator will clinically evaluate the patient and the patient will complete self assessment documents, Oswestry Disability Index, Quality of Life questionnaires and a surgery satisfaction survey, e.g., very satisfied, satisfied, somewhat unsatisfied, or very unsatisfied with the surgery. Fusion status will be evaluated radiographically at each visit using plain films. CT scans at 12 months will be evaluated by an independent radiologist. Complication data will be recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

The patient can be included in the study if all of the following criteria are met;

1. is at least 18 years of age and skeletally mature
2. must have symptomatic spinal stenosis and/or spondylolisthesis or degenerative disc disease (DDD) at one or two adjacent levels from L2-S1 requiring a fusion
3. must have completed a minimum of three months of unsuccessful conservative, non-operative care
4. must have discogenic back pain with or without leg pain
5. DDD must be confirmed by MRI or CT scans followed by discography (if necessary)
6. must score at least 40 points on the Oswestry Disability Index
7. must score at least a 4 on a 10 cm Visual Analog Scale for back pain
8. must be able to comply with the protocol"s follow-up schedule
9. must understand and sign the informed consent document

Exclusion Criteria:

The patient must not exhibit any of the following criteria;

1. symptomatic at more than two levels
2. previous fusion surgery at any lumbar level with or without instrumentation (prior discectomy, laminotomy, laminectomy or nucleolysis at the operative (involved) level > 6 months is permitted)
3. more than 50% spondylolisthesis
4. lumbar scoliosis greater than 11 degrees
5. osteoporosis*, osteopenia, osteomalacia, Paget"s disease or metabolic bone disease.
6. spinal tumors
7. active arachnoiditis Pioneer Surgical Technology Confidential nanOss Bioactive Post Marketing Clinical Study: March 11, 2010 Page 8
8. fractures of the epiphyseal plate or fractures for which stabilization of the fracture is not possible.
9. Impaired calcium metabolism
10. active infection or surgical site infection
11. rheumatoid arthritis or other autoimmune disease
12. chronic steroid use (used steroids for one month within the last 6 months) or any medical condition that requires treatment with drugs known to interfere with bone healing
13. systemic disease such as AIDS, HIV, hepatitis (active), tuberculosis
14. morbid obesity defined as body mass index (BMI) >40 or a weight more than 100 lbs over ideal body weight
15. smokers unless the patient agrees to quit at least 2 weeks prior to and for the duration of the study, confirmed by a carboxyhemoglobin test prior to surgery
16. psychosocial disorders that would preclude accurate evaluation or has a history of substance abuse
17. active malignancy except non-melanoma skin cancer; history of any invasive malignancy unless treated and in remission for at least five years
18. documented allergies to porcine collagen or titanium
19. pregnancy, or interested in becoming pregnant in the next four years
20. participation in another investigational study within 30 days *Osteoporosis will be assessed at the time of the preoperative evaluation based on the patient"s history, physical examination and review of the radiographic evaluations. All patients at risk for osteoporosis must obtain a DEXA scan of the spine and hip to determine if the patient has severe osteoporosis. The definition of a patient at risk used by the National Osteoporosis Foundation includes the following: i. Premature menopause (< 45 years) ii. Prolonged amenorrhea (> one year) iii. Maternal history of hip fracture iv. Primary hyperparathyroidism or hyperthyroidism v. Chronic renal failure vi. Previous fragility fractures, particularly of the hip, spine or wrist vii. Patients who have ever taken corticosteroids in doses >7.5 mg/day for one year or more. Patients will be excluded if their bone mineral density (BMD) in the spine or hip is more than 1.0 standard deviation (SD) below the mean of normal adults in the presence of one or more fragility fractures indicating severe osteoporosis. If severe osteoporosis is diagnosed, the patient must be excluded from the investigational study. If the patient has osteoporosis or osteopenia, they may be included in the study if he or she meets the rest of the inclusion and exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Spinal fusion | 12 months
  1. Bridging trabecular bone
  2. Less than 3mm of translational motion
  3. Less than 5mm of angular motion

SECONDARY OUTCOMES:
Improvement in Oswestry Disability Index score | 12 months
Improvement in VAS pain scores | 12 months
Improvement in Quality of Life scores | 12 months
Decrease in medication usage | 12 months
Patient returning to work | 12 months
Patient satisfaction (surgery satisfaction survey, e.g., very satisfied, satisfied, somewhat unsatisfied, or very unsatisfied with the surgery) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Songer, MD, Principal Investigator — Advanced Center for Orthopedics
Locations (7):
- United States (7):
  - Tower Orthopaedics & Neurosurgical Spine Institute, Beverly Hills, California
  - Scripps Memorial Hospital Neurosurgery, La Jolla, California
  - Northwestern Medical Facility, Chicago, Illinois
  - Advanced Center for Orthopedics, Marquette, Michigan
  - St. Johns Spine and Pain Clinic, Springfield, Missouri
  - Medical University of South Carolina Neurology, Charleston, South Carolina
  - Milwaukee Spinal Specialists, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No